CLINICAL TRIAL: NCT03441321
Title: Randomized Trial of a Social Media-Delivered Intervention
Brief Title: Social-Media Intervention in Reducing Tanning in High-Risk Tanners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jerod L Stapleton, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jerod L Stapleton, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 56153; NCI-2018-00168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000184; 131704 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); R01CA218068 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Health Status Unknown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (focusing on tanning and healthy body image) (Experimental): Participants periodically read the content on the study-specific private and hidden Facebook group related to living a healthy lifestyle including avoiding tanning and excessive ultraviolet exposure, managing stress, healthy eating, promoting physically active lifestyles, and promoting a healthy body image, and participate in the group by providing reactions, commenting on the posts, or by sharing study relevant information within the group for 8 weeks.
  Interventions: Other: Lifestyle and Values Intervention; Other: Survey Administration
- Group II (focusing on other health topics) (Active Comparator): Participants participate in private and hidden Facebook groups that utilize content from the intervention content library related to other health topics of interest (e.g., physical activity, healthy eating, alcohol misuse prevention, stress reduction, sleep) for 8 weeks.
  Interventions: Other: Lifestyle Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Lifestyle and Values Intervention — Participate in Facebook group focusing on avoiding tanning and promoting healthy body image
  Arms: Group I (focusing on tanning and healthy body image)
Other: Lifestyle Intervention — Participate in Facebook group focusing on other health topics
  Arms: Group II (focusing on other health topics)
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well social-media intervention works in reducing tanning in high-risk indoor and outdoor tanners. Social-media intervention delivered via Facebook may help to promote healthy behaviors, positive body image, and to understand young women's perception of a social media campaign.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a randomized control trial to examine the efficacy of the intervention versus (vs.) a Facebook-delivered control group on reducing tanning behavior among high-risk indoor and outdoor tanners.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants periodically read the content on the study-specific secret Facebook group related to living a healthy lifestyle including avoiding tanning and excessive ultraviolet exposure, managing stress, healthy eating, promoting physically active lifestyles, and promoting a healthy body image, and participate in the group by providing reactions, commenting on the posts, or by sharing study relevant information within the group for 8 weeks.

GROUP II: Participants participate in secret Facebook groups that utilize content from the intervention content library related to other health topics of interest (e.g., physical activity, healthy eating, alcohol misuse prevention, stress reduction, sleep) for 8 weeks.

After completion of study, patients are followed up at 3, 8, and 18 months post baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* High-risk indoor or outdoor tanner (defined as using an indoor tanning bed or intentionally tanning outdoors at least 10 times in the previous 12 months)
* Use of Facebook at least 4 times per week

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 407 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Number of indoor or outdoor tanning sessions assessed using surveys | At 8 months
  Multilevel models (e.g., random coefficient) will be used to test the primary study hypothesis that participants who received the intervention will report less combined indoor and outdoor tanning behavior at a 8-month follow-up compared to those who received the control. If necessary, sensitivity analyses may control for individual-level covariates.

SECONDARY OUTCOMES:
Indoor and outdoor tanning behavior assessed using surveys | At 18 months
  Multilevel models (e.g., random coefficient) will be used. If necessary, sensitivity analyses may control for individual-level covariates.
Skin burns from indoor and outdoor tanning assessed using surveys | At 8 months
  Multilevel models (e.g., random coefficient) will be used. If necessary, sensitivity analyses may control for individual-level covariates.
Tanning intentions assessed using surveys | At 8 months
  Multilevel models (e.g., random coefficient) will be used. If necessary, sensitivity analyses may control for individual-level covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Jerod Stapleton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stapleton JL, Manne SL, Pagoto SL, Leip A, Greene K, Hillhouse JJ, Merritt AS, Shelton BJ. A Social Media-Delivered Melanoma Prevention Program for Young Women Engaged in Frequent UV Tanning: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 19;13:e56562. doi: 10.2196/56562. PMID 38502173

DOCUMENTS (1):
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT03441321/ICF_000.pdf